CLINICAL TRIAL: NCT04066569
Title: Reproducibility and Utility of Growth Hormone Inhibition by Oral Glucose Tolerance Test for the Diagnosis of Acromegaly
Brief Title: Reproducibility and Utility of OGTT in Acromegaly
Acronym: ACROTEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P170917J
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Acromegaly
Keywords: Diagnostic test; Growth hormone; oral glucose tolerance test
MeSH Terms: conditions — Acromegaly | interventions — Glucose; Aspartame

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OGTT Tests and Placebo Test (Active Comparator): Patients with acromegaly
  Interventions: Other: Performed 3 diagnostic tests (2 OGTT tests with 75 g of Glucose and 1 placebo test with 375 mg of Aspartam
- OGTT Tests (Active Comparator): age and sex matched healthy volunteers
  Interventions: Other: Performed 2 diagnostic tests (2 OGTT tests with 75g of Glucose)

INTERVENTIONS:
Other: Performed 3 diagnostic tests (2 OGTT tests with 75 g of Glucose and 1 placebo test with 375 mg of Aspartam — After inclusion, the study will include the sequential realization of 3 dynamic GH secretion tests, separated by a period of 24 hours to 30 days. Each subject will have two OGTT tests (oral administration of 75 g of glucose in 200 mL of water) and a placebo test (oral administration of 375 mg of aspartame in 200 mL of water). The order of the three tests (2 OGTT and 1 placebo) in acromegalic patients will be randomized.
  The tests will be performed under the same conditions
  Arms: OGTT Tests and Placebo Test
Other: Performed 2 diagnostic tests (2 OGTT tests with 75g of Glucose) — After inclusion, the study will include the sequential realization of 2 dynamic GH secretion tests, separated by a period of 24 hours to 30 days. Each subject will have two OGTT tests (oral administration of 75 g of glucose in 200 mL of water).
  The tests will be performed under the same conditions (fasting, semi-recumbent position, start of the test at 9 am) and will include a measurement of blood glucose, GH, insulinemia at -15, 0, 30, 60, 90, 120 min after ingestion of glucose or placebo.
  Arms: OGTT Tests

SUMMARY:
Prospective study of reproducibility and utility of growth hormone inhibition by oral glucose tolerance test for the diagnosis of acromegaly, in acromegalic and non-acromegalic subjects, with a randomized double-blind crossover over placebo arm in the group of acromegalic patients

DETAILED DESCRIPTION:
Rational: The initial step of biological diagnosis of acromegaly is based on assessment of IGF-I. According to current recommendations, the diagnosis must be confirmed by an oral glucose tolerance test (OGTT) to show that there is no growth hormone (GH) decrease lower than 1 μg/L (Katznelson , et al., 2014).

Reproducibility of GH suppression by the OGTT has never been evaluated in either acromegalic or healthy subjects, although it is essential to determine the reliability of this test. Spontaneous fluctuations in GH in acromegaly could significantly influence the response of GH to the OGTT and cause low reproducibility of the test in this population. In particular, this reliability could be different according to the typical or moderate clinical presentation because of the persistence of a residual ultradian rhythm of GH secretion.

The usefulness of oral glucose loading and the resulting hyperglycemia (which may limit GH secretion) has never been compared to an appropriate placebo (aspartame, at a dose equivalent to 75 g glucose), which does not cause hyperglycemia. Ingestion of 75 g of glucose is often responsible for nausea and vomiting. More rarely, the drop in blood glucose reactive to hyper insulinemia at the end of the test, can be the cause of discomfort.

Primary objective: To determine the reproducibility of the GH response to OGTT in acromegaly by studying, in subjects with acromegaly, changes in GH concentration within 2 hours after oral administration of 75 g of glucose at 2 repeated tests in the same subject.

Secondary objectives:

1. To analyze the reproducibility of the GH response to the OGTT as a function of the severity of acromegaly ("typical" form, "intermediate" form of acromegaly) and in a group of non-acromegalic subjects.
2. To evaluate the diagnostic value (utility) of OGTT in acromegaly by comparing, in subjects with acromegaly, the response of GH to oral administration of 75 g of glucose (OGTT) and 375 mg of aspartame (placebo).
3. Evaluate OGTT-stimulated insulin secretion in acromegalic and non-acromegalic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Acromegalic subjects
* Men or women, adults ≤ 85 years, with hypersecretion of GH proven by the following criteria:

  * High IGF-I compared to age and sex standards (Variety study, Chanson et al., 2016)
  * and basal GH concentrations > 0.4 μg / L (Katznelson, et al., 2014) and somatotropic pituitary adenoma operated on or planned to be operated on. It may be patients whose acromegaly has just been discovered and not yet treated (de novo patients) for whom a surgical treatment is envisaged within 6 months after inclusion or acromegalic patients already operated on a pituitary adenoma whose acromegaly is not controlled by surgery. A histological confirmation of a somatotropic pituitary adenoma will be obtained either before inclusion in the study (subjects already operated) or after inclusion ("de novo" subjects) in order to have a sufficient level of proof of the diagnosis of acromegaly, especially in the "intermediate" forms.
* Medically treated patients who decide to discontinue treatment (in order to reassess the progression of the disease, or at the time of a change), will be eligible after more than 3 months of discontinuation of the drug treatment.
* In women on estrogen / progestin contraception, this should be kept unchanged throughout the study. In the absence of estrogen / progestin contraception, exploration will be done in the follicular phase.

Non-acromegalic subjects:

* Men or women, adults ≤ 85 years
* Subjects defined by a concentration of IGF-I below 100% of the upper limit of normal, matched for sex and age (± 5 years) to acromegalic patients.
* Normal blood pressure measured by an electronic tensiometer validated after 5 min resting in supine position <140/90 mmHg on 3 consecutive measurements
* Biological assessment (hematological and biochemical blood tests, urine analysis) within the limits of normal or clinically acceptable. Normal EKG.
* ECG 12 leads without particularity.
* Affiliation to a social security scheme
* At the women on estrogen-progestative contraception, this one should be kept unchanged throughout the study. In the absence of estrogen-progestative contraception,the exploration will be done in the follicular phase.
* Signed informed consent.

Exclusion Criteria:

For both groups:

* Pregnant or breastfeeding women
* Acute systemic diseases
* Pathologies likely to affect digestive absorption
* Taking prohibited treatments (see section 7.3)
* History of hypersensitivity to aspartame (edema of Quincke, Urticaria ..)
* Donation of blood in the 3 months preceding the study
* People in the exclusion period on the national file people suitable for research involving the human person
* Refusal or linguistic or psychic incapacity to sign informed consent
* Subject unable to submit to the constraints of the protocol (for example, non-cooperating, unable to return to follow-up visits and probably unable to finish the study)
* Major under guardianship
* Major under curatorship
* People with phenylketonuria
* Person with digestive intolerance to glucose /galactose, digestive labsorption syndrome of glucose / galactose.

For the group of acromegalic patients:

* acromegalic patients with diabetes mellitus treated with insulin
* Acromegalic patients under medical treatment of their acromegaly somatostatin analogues, pegvisomant), or patients in whom this treatment has been suspended for less than 3 months at the time of the selection.
* Acromegalic patients who have been treated with radiotherapy.

For the group of non-acromegalic subjects:

- Chronic systemic diseases likely to influence the secretion of GH like diabetes sweetness, severe obesity (BMI> 35 kg / m2), inadequate renal (creatinine clearance <60 mL / min), disease hypothalamic-pituitary, epilepsy, antecedents Hepatocellular insufficiency and insufficiency cardiac, progressive cancer.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Compare Nadir GH concentration in μg/L obtained in two OGTT in the same subject with acromegaly | The two test will be separated by the preiod of 24h - 30 days
  GH will be measured by an immunometric chemiluminescent assay on an Immulite 2000XPi (Siemens Healthcare Diagnostics, Erlangen, Germany) on venous blood samples at -15 min, 0 min, 30 min, 60 min, 90 min, 120 min after ingestion of 75g of glucose

SECONDARY OUTCOMES:
Severity of acromegaly ("typical" form, "intermediate" form of acromegaly) | The two test will be separated by the preiod of 24h - 30 days
  "Typical" form of acromegaly defined by an IGF-I concentration> 200% of the upper limit of normal, in the presence of a somatotropic pituitary adenoma
  • moderate or "intermediate" form of acromegaly defined by an IGF-I concentration value between 100% and 200% of the upper limit of normal, in the presence of a somatotropic pituitary adenoma. The IGF-I reference values determined by sex and age in the "Variety" study will be used for this classification
Nadir GH in mIU / L (conversion 1 μg / L = 3 mIU / L) obtained in the two OGTT tests and the placebo (aspartame) test repeated in the same subject (acromegalic and non acromegalic) | Each test will be separated by the preiod of 24h - 30 days
  Nadir GH in ug/L obtained in the two OGTT tests and the placebo (aspartame) test repeated in the same subject. GH will be measured by an immunometric chemiluminescent assay on an Immulite 2000XPi (Siemens Healthcare Diagnostics, Erlangen, Germany) on venous blood samples at -15 min, 0 min , 30 min , 60 min , 90 min , 120 min after ingestion of 75g of glucose / 375g of aspartame
Peak glucose level in both OGTT and placebo tests | Each test will be separated by the preiod of 24h - 30 days
  Verification of hyperglycemia induced or not depending on the product administered

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No